CLINICAL TRIAL: NCT01365026
Title: Feasibility and Effectiveness of Innovative Programs for Health Promotion in Primary Care: The 'Prescribe Healthy Life' Project (PVS)
Brief Title: PVS: Innovative Programs For Healthy Lifestyle Promotion in Primary Care: 'Prescribe Healthy Life'
Acronym: PVS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Gonzalo Grandes, MD, MS Epidemiology, Basque Health Service
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PS09/01461; 2014111076 (Other Grant/Funding Number: Basque Health Department); PI13/00573 (Other Grant/Funding Number: Carlos III Institute of Health, Spanish Ministry of Health); RD12/0005/0010 (Other Grant/Funding Number: Carlos III Institute of Health, Spanish Ministry of Health)
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Health Promotion; Health Education; Patient Education; Counseling; Behavior Therapy; Health Behavior
Keywords: Healthy Lifestyle; Health promotion; Counselling; Action Plan; Primary Health Care
MeSH Terms: conditions — Health Education; Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PVS intervention (Experimental)
  Interventions: Behavioral: PVS: Programa de Vida Saludable
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: PVS: Programa de Vida Saludable — Lifestyle counseling and prescription
  Arms: PVS intervention

SUMMARY:
The potential health gains from healthy lifestyles are very well-known, what is still not known is how to help people to adopt these lifestyles, by means of brief interventions feasible in routine general practice. This study was designed to explore the feasibility and efficacy of innovative implementation strategies for the promotion physical activity, diet and smoking abstinence in primary care. The investigators hypothesize that collegiate planning between practitioners, researchers and managers, with a socio-ecological perspective and taking into account the real context of collaborating centers, will guarantee the sustainability and effectiveness of these programs.

DETAILED DESCRIPTION:
BACKGROUND: Primary health care (PHC) services have special opportunities for healthy lifestyles promotion. Yet, despite its potential impact health promotion is not widespread and the results obtained are limited.

OBJECTIVE: To explore the feasibility and efficacy of an implementation strategy for optimizing the promotion of physical activity, diet and smoking abstinence in PHC. The strategy is innovative for its collegiate planning between practitioners, researchers and managers, with a socio-ecological perspective and taking into account the real context of collaborating centers.

DESIGN AND LOCATION: quasi-experimental hybrid implementation-effectiveness trial, conducted in 6 PHC centers (20 practices in 3 intervention centers and 21 in 3 control centers), with the collaboration of the majority of primary care professionals within each center, and the participation of 4017 attendees randomly selected from the target population. INTERVENTION CENTRES: Each of the intervention centers will be exposed to the PVS multicomponent implementation strategy, including training, information and communication electronic tools integrated into the electronic clinical record (ECR), local leadership, creation of a community of practice, practice facilitation, and audit and feed-back for the implementation of an intervention program to promote multiple healthy lifestyles (physical activity, healthy diet, and smoking cessation), based on the 5A's (Ask, Advise, Agree, Assist and Arrange follow-up), and modeled by professionals in each intervention center, according to their organizational context and available community resources and agents.

CONTROL CENTRES: will receive the same training and dissemination of clinical guidelines, electronic support tools integrated into the ECR, audit and feed-back.

MEASUREMENTS: Programs' implementation will be evaluated in terms of reach, adoption, implementation and acceptability by PHC staff, following the RE-AIM framework. PHC attendees will be followed with 2 repeated measurements at baseline, and 6 months to estimate change in patients' adoption of the minimum recommended level of healthy lifestyles.

ANALYSIS: the investigators will compare the implementation rate of health promotion activities in intervention and control centers, the proportion of users exposed to the 5 A's and the observed change in users' healthy lifestyles. Centers with different intensities of actual implementation will be compared to explore characteristics associated with implementation and the interaction between implementation strategies and clinical effectiveness of the intervention programs.

ELIGIBILITY:
Inclusion Criteria:

* primary care attendees not meeting at least one of the healthy lifestyles recommendations
* 10 to 80 years old

Exclusion Criteria:

* psychotic mental disorders
* brain degenerative disorders
* mental retardation
* cognitive impairment
* dementia
* end of life

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4017 (Estimated)
Dates: Start 2016-01-06 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Health propmotion clinical practice change | 12 months
  Rates and proportion of primary care attendees exposed to the 5 A's
Adoption by primary care attendees of the minimum recommended levels of physical activity, fruits and vegetable consumption and smoking abstinence | 6 months
  Change in at least one and number of modified lifestyle behaviors

SECONDARY OUTCOMES:
Efficiency of healthy lifestyle prescription | 6 months
  Costs and utility of the prescription of healthy behabior change plan

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Grandes, MD, MS, Principal Investigator — Basque Health Service
Locations (1):
- Primary Care Research Unit of Bizkaia, Bilbao, Spain

REFERENCES:
- [Background] Sanchez A, Grandes G, Cortada JM, Pombo H, Balague L, Calderon C. Modelling innovative interventions for optimising healthy lifestyle promotion in primary health care: "prescribe Vida Saludable" phase I research protocol. BMC Health Serv Res. 2009 Jun 18;9:103. doi: 10.1186/1472-6963-9-103. PMID 19534832
- [Background] Grandes G, Sanchez A, Cortada JM, Balague L, Calderon C, Arrazola A, Vergara I, Millan E; Prescribe Vida Saludable group. Is integration of healthy lifestyle promotion into primary care feasible? Discussion and consensus sessions between clinicians and researchers. BMC Health Serv Res. 2008 Oct 14;8:213. doi: 10.1186/1472-6963-8-213. PMID 18854033
- [Background] Grandes G, Sanchez A, Sanchez-Pinilla RO, Torcal J, Montoya I, Lizarraga K, Serra J; PEPAF Group. Effectiveness of physical activity advice and prescription by physicians in routine primary care: a cluster randomized trial. Arch Intern Med. 2009 Apr 13;169(7):694-701. doi: 10.1001/archinternmed.2009.23. PMID 19364999
- [Background] Grandes G, Sanchez A, Torcal J, Sanchez-Pinilla RO, Lizarraga K, Serra J; PEPAF Group. Targeting physical activity promotion in general practice: characteristics of inactive patients and willingness to change. BMC Public Health. 2008 May 22;8:172. doi: 10.1186/1471-2458-8-172. PMID 18498623
- [Background] Zuazagoitia A, Montoya I, Grandes G, Arietaleanizbeascoa MS, Arce V, Martinez V, Sanchez M, Sanchez A. Reliability and validity of the 7-day Physical Activity Recall interview in a Spanish population. Eur J Sport Sci. 2014;14 Suppl 1:S361-8. doi: 10.1080/17461391.2012.705332. Epub 2012 Jul 25. PMID 24444230
- [Background] Sanchez A, Grandes G, Ortega Sanchez-Pinilla R, Torcal J, Montoya I; PEPAF Group. Predictors of long-term change of a physical activity promotion programme in primary care. BMC Public Health. 2014 Feb 4;14:108. doi: 10.1186/1471-2458-14-108. PMID 24491081
- [Background] Sanchez A, Bully P, Martinez C, Grandes G. Effectiveness of physical activity promotion interventions in primary care: A review of reviews. Prev Med. 2015 Jul;76 Suppl:S56-67. doi: 10.1016/j.ypmed.2014.09.012. Epub 2014 Sep 26. PMID 25263343
- [Background] Bully P, Sanchez A, Zabaleta-del-Olmo E, Pombo H, Grandes G. Evidence from interventions based on theoretical models for lifestyle modification (physical activity, diet, alcohol and tobacco use) in primary care settings: A systematic review. Prev Med. 2015 Jul;76 Suppl:S76-93. doi: 10.1016/j.ypmed.2014.12.020. Epub 2015 Jan 5. PMID 25572619
- [Background] Sanchez A, Silvestre C, Campo N, Grandes G; PreDE research group. Type-2 diabetes primary prevention program implemented in routine primary care: a process evaluation study. Trials. 2016 May 20;17(1):254. doi: 10.1186/s13063-016-1379-0. PMID 27206733
- [Background] Bully P, Sanchez A, Grandes G, Pombo H, Arietalenizbeaskoa MS, Arce V, Martinez C; PVS Group. Metric properties of the "prescribe healthy life" screening questionnaire to detect healthy behaviors: a cross-sectional pilot study. BMC Public Health. 2016 Dec 7;16(1):1228. doi: 10.1186/s12889-016-3898-8. PMID 27923356